CLINICAL TRIAL: NCT01479036
Title: Phase Ⅲ Trial of Neoadjuvant Recombinant Human Endostatin, Docetaxel and Epirubicin as First-Line Therapy in Patients With Breast Cancer
Brief Title: Trial of Neoadjuvant Endostar, Docetaxel and Epirubicin for Patients With Breast Cancer
Acronym: CBCRT01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Endostar B-02; CBCRT01 (Other Grant/Funding Number: NNSF of China (No. 81172510, 30872514))
Record Dates: First submitted 2011-10-26; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant chemotherapy; recombinant human endostatin (endostar); docetaxel; epirubicin
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin; Endostatins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- docetaxel and epirubicin (Active Comparator): DE chemotherapy alone
  Interventions: Drug: docetaxel and epirubicin
- docetaxel and epirubicin plus endostatin (Experimental): chemotherapy plus endostatin
  Interventions: Drug: docetaxel and epirubicin plus endostatin

INTERVENTIONS:
Drug: docetaxel and epirubicin — docetaxel 75mg/m2, IV (in the vein) on day 1 of each 21 day cycle; epirubicin 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle, totally 3 cycles
  Other Names: Docetaxel, Sanofi-Aventis; Epirubicin, Pfizer
  Arms: docetaxel and epirubicin
Drug: docetaxel and epirubicin plus endostatin — docetaxel 75mg/m2, IV (in the vein) on day 1 of each 21 day cycle; epirubicin 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle; endostatin 7.5mg/m2, IV (in the vein) on 1st to 14th days of each 21 day cycle; every 3 weeks, totally 3 cycles
  Other Names: Endostatin, Simcere-Medgenn (No. S20050088)
  Arms: docetaxel and epirubicin plus endostatin

SUMMARY:
This study was designed to determine the efficacy and safety of neoadjuvant docetaxel and epirubicin (DE) with or without human recombinant endostatin (endostar) for breast cancer patients. The hypothesis of this protocol is that a combined angiogenesis inhibiting therapy to chemotherapy could further benefit breast cancer patients.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, controlled phase Ⅲ clinical trial. A total of 800 patients with core-biopsy confirmed breast cancer, stage ⅡA to ⅢC, and to be treated with neoadjuvant systemic therapy are eligible for entry into this study. Patients will be allocated randomly to two groups to receive either 3 cycles of neoadjuvant DE and endostar or 3 cycles of neoadjuvant DE. All cases receive mammography, contrast-enhanced ultrasound (CEUS), magnetic resonance angiography (MRA), and positron emission tomography (PET) scanning pre- and post-neoadjuvant therapy, and then undergo surgical resection. The primary endpoint is clinical/pathological response. The clinical response will be evaluated according to RECIST criteria. The parameters of tumor metabolism and blood supply, as demonstrated by PET, MRA and CEUS, will be collected and analysed. The secondary endpoint is (1) the number of participants with adverse events, (2) quality of life scores, and (3) the number of adverse events reported during neoadjuvant therapy. In addition, the role of mammography, CEUS, MRA and PET for response evaluation, as well as the angiogenic profile and biological information involved in tumor response will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer (core needle biopsy for breast cancer diagnosis and fine needle aspiration for lymph node metastasis diagnosis)
* Stage ⅡA-ⅢC
* Age 18-70
* ECOG performance status 0-2
* No evidence of distant metastasis
* No previous therapy
* Normal hematologic function
* left ventricular ejection fraction greater than 50 percent
* No abnormality of renal or liver function
* Written informed consent

Exclusion Criteria:

* With allergic constitution or possible allergic reflection to drugs to be used in this study
* Any concurrent uncontrolled medical or psychiatric disorder
* History of severe heart diseases, including congestive heart failure, unstable angina, uncontrolled arrhythmia, myocardial infarction, uncontrolled high blood pressure, or heart valve disease.
* History of bleeding diathesis
* Being pregnant or nursing

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2011-10; Primary Completion 2014-12 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Clinical/pathological response | 3 years
  The clincial response will be evaluated according to RECIST criteria. The parameters of tumor metabolism and blood supply, as demonstrated by PET, MRA and CEUS, will be collected and analysed.

SECONDARY OUTCOMES:
Number of participants with adverse events | 3 years
  The number of participants with adverse events will be recorded and analysed.
Quality of life | 3 years
  Quality of life is scored using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life of Questionnaire (QLQ30) at study entry and prior to surgery.
Number of adverse events reported during neoadjuvant therapy | 3 years
  The adverse events during neoadjuvant therapy will be graded using the National Cancer Institute Common Toxicity Criteria (NCI CTC) version 2.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jianghao Chen, MD, PhD, Principal Investigator — Xijing Hospital; Ling Wang, MD, Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] In our previous phase Ⅱ trial (NCT00604435), the combination of rh-endostatin with docetaxel and epirubicin chemotherapy resulted in a higher objective response rate without increased toxicity in breast cancer patients, as compared with chemotherapy alone. Our results have been accepted to report as General Poster in ASCO's 47th Annual Meeting in 2011. Wang L, Chen JH, Yao Q, et al. Neoadjuvant rh-endostatin, docetaxel and epirubicin for breast cancer: efficacy and safety in a prospective, randomized, phase II study. 2011 ASCO Annual Meeting Proceedings, J Clin Oncol 2011; 29(15s): 112s.
- [Derived] Chen J, Yao Q, Huang M, Wang B, Zhang J, Wang T, Ming Y, Zhou X, Jia Q, Huan Y, Wang J, Wang L. A randomized Phase III trial of neoadjuvant recombinant human endostatin, docetaxel and epirubicin as first-line therapy for patients with breast cancer (CBCRT01). Int J Cancer. 2018 May 15;142(10):2130-2138. doi: 10.1002/ijc.31217. Epub 2017 Dec 23. PMID 29238974